CLINICAL TRIAL: NCT06520293
Title: Effects of a Single Oral Dose of Sweet Protein Sweelin® on Blood Glucose and Insulin Levels in Healthy Adults: a Crossover, Double Blinded Clinical Trial
Brief Title: Effects of a Single Oral Dose of Sweet Protein Sweelin® on Blood Glucose and Insulin Levels in Healthy Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amai Proteins (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: SWEELIN01
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Beverage containing Serendipity Berry Sweet Protein (Experimental): Single dose of 400 ml beverage containing Serendipity Berry Sweet Protein to be consumed in less than 15 minutes. The beverage will be at a similar sweet potency as 75 grams glucose.
  Interventions: Other: Sweet Beverage
- Beverage containing glucose (Other): Single dose of 400 ml beverage containing 75 grams glucose to be consumed in less than 15 minutes.
  Interventions: Other: Sweet Beverage
- Beverage containing Stevia (Other): Single dose of 400 ml beverage containing Stevia to be consumed in less than 15 minutes. The beverage will be at a similar sweet potency as 75 grams glucose.
  Interventions: Other: Sweet Beverage

INTERVENTIONS:
Other: Sweet Beverage — A beverage containing different sweet ingredients.

SUMMARY:
The study aims to evaluate, for the first time, the post-prandial effects of a single oral administration of Serendipity Berry Sweet Protein sweelin® compared to glucose and stevia, as a commercial sweetener, in healthy adults. The study design is a single center, randomized, crossover study.

Each subject will receive a single oral dose of sweelin® compared with an equivalently sweet dose of glucose and stevia dissolved in a water beverage with flavor.

The advantage of a crossover design is that it will allow to compare the blood glucose and insulin levels of each subject to his baseline in every test beverage, and to remove the inter-subject variability. The post-prandial effects will be monitored with multiple blood sampling up to 120 minutes post dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects
2. Age 18-70 years
3. BMI between 18.0 and 33.0 calculated as Weight (Kg)/Height (m2).
4. Stable weight in the last 3 months (+/-5kg).
5. Subjects must be able to adhere to the visit schedule and protocol requirements and be available to complete the study.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Subjects with a significant allergic response or history of food allergies deemed clinically significant or exclusionary for the study.
3. Diabetes mellitus or use of medications affecting glucose metabolism.
4. Subjects with any gastrointestinal disease which may affect absorption
5. Subjects with any acute medical situation (e.g. acute infection) within 48 hours of study start, which is considered of significance by the Principal Investigator.
6. Subjects which have undergone major surgery in the last 3 months.
7. Subjects who are non-cooperative or unwilling to sign the consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Blood glucose incremental area under the curve (iAUC) | 120 minutes after single oral dose administration
  To monitor blood glucose incremental area under the curve (iAUC) response of sweelin® in healthy adult subjects, following a single oral administration, in comparison to glucose and stevia.

SECONDARY OUTCOMES:
Insulin incremental area under the curve (iAUC) | 120 minutes after single oral dose administration
  To monitor blood insulin incremental area under the curve (iAUC) response of sweelin®, following a single oral administration, in comparison to glucose and stevia.

CONTACTS AND LOCATIONS:
Overall Officials: David Zeltser, Prof., Principal Investigator — Tel-Aviv Sourasky Medical Center

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: within one year post study completion
Access Criteria: Interested researchers must submit a formal data access request via email to the sponsor- Amai Proteins yael.lifshitz@amaiproteins.com